CLINICAL TRIAL: NCT03631927
Title: Indian Intensive Care Case Mix and Practice Patterns Study - II
Brief Title: Second Survey of Intensive Care in India
Acronym: INDICAPS-II
Status: Completed | Type: Observational
Sponsor: Indian Society of Critical Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: INDICAPS2
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Critical Illness
Keywords: critical care unit
MeSH Terms: conditions — Critical Illness | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients admitted to participating ICUs on the specified dates
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
INDICAPS was the first large scale, multicentre survey launched by the ISCCM. The aim was to gather information about ICUs, organizational characteristics, patient casemix, the types and severity of illness, monitoring and therapeutic modalities used, types of infections, and other such data. This was performed between July 2010 and April 2011 and published in 2016.[1] Over the last 8 years, there has been a significant difference in the delivery of intensive care services, critical care education, socioeconomic indicators, antibiotic resistance patterns and other aspects of practices in Indian ICUs. It is therefore necessary to revisit and resurvey the current trends in intensive care practices in India, and to reflect the vast spectrum of critical care illness, services and practices.

Similar to INDICAPS, which was a point-prevalence study of all patients present in the ICU on four different days over a one-year period, INDICAPS II will record data of all patients admitted to the ICU on 4 different days.

DETAILED DESCRIPTION:
INDICAPS II will record data of all patients admitted to the ICU on 4 different days (August 23, 2018; October 25, 2018; December 13, 2018; April 11, 2019) in a cross-sectional design. Data collection includes:

1. On admission: demographic characteristics, comorbidities, source of admission, primary and secondary admission diagnoses,
2. Baseline data (on the study day), including parameters used to calculate SAPS II score and SOFA score and infections,
3. Information on monitoring modalities, mechanical ventilation, nutrition, fluid therapy, other routine ICU practices

c. Outcome at ICU and hospital discharge d. Organisation of ICU services

ELIGIBILITY:
Inclusion Criteria:

* All patients present in the ICU on August 23, 2018; October 25, 2018; December 13, 2018; April 11, 2019

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients present in the ICU on August 23, 2018; October 25, 2018; December 13, 2018; April 11, 2019
Sampling Method: Non-Probability Sample
Enrollment: 5094 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jigeeshu V Divatia, MD, FCCM, Study Chair — Tata Memorial Hospital
Locations (108):
- India (108):
  - Nri Medical College & General Hospital, Guntur, Andhra Pradesh
  - CARE Hospitals, Visakhapatnam, Andhra Pradesh
  - Sevenhills Hospital, Visakhapatnam, Andhra Pradesh
  - Nemcare Hospital, Guwahati, Assam
  - Apollo hospitals, Guwahati, Assam
  - Ayursundra superspecialty Hospital, Guwahati, Assam
  - Paras Hmri Hospital, Patna, Bihar
  - All India Institute of Medical Sciences,Patna, Patna, Bihar
  - Hcg Hospitals, Ahmedabad, Gujarat
  - Sterling hospital, Ahmedabad, Gujarat
  - CIMS Hospital, Ahmedabad, Gujarat
  - Apollo Hospital International Ltd, Ahmedabad, Gujarat
  - Shree Krishna Hospital, Anand, Gujarat
  - Mangalam hospital, Morvi, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Synergy Superspeciality Hospital, Rajkot, Gujarat
  - Spandan Multispeciality Hospital, Vadodara, Gujarat
  - GMERS Gotri Medical college, Vadodara, Gujarat
  - Dhiraj hospital SBKSMIRC, Vadodara, Gujarat
  - Asian Institute of Medical Sciences, Faridabad, Haryana
  - Artemis Health Institute, Gurgaon, Haryana
  - Medanta - The Medicity, Gurgaon, Haryana
  - Medanta The Medicity, Gurgaon, Haryana
  - ASCOMS, Jammu, Jammu and Kashmir
  - St John's Medical College Hospital, Bangalore, Karnataka
  - Sri Shankara Cancer Hospital and Research Center, Bengaluru, Karnataka
  - Manipal hospital Whitefield, Bengaluru, Karnataka
  - Narayana Hrudayalaya, Bengaluru, Karnataka
  - Shri Ganpatlal Agarwal Memorial Ayush Multi-specialty Hospital and Research Center, Vijayapura, Karnataka
  - Aster Medcity, Kochi, Kerala
  - Holy Family Hospital, Thodupuzha, Kerala
  - Chirayu Medical College and Hospital Bhopal, Bhopal, Madhya Pradesh
  - Choithram hospital and research centre, Indore, Madhya Pradesh
  - Chirayu hospital, Rewa, Madhya Pradesh
  - Sagar shree hospital, Sāgar, Madhya Pradesh
  - Ozone Multispeciality Hospital, Akola, Maharashtra
  - MGM MCRI and Hospital, Aurangabad, Maharashtra
  - BKL Walawalkar Rural Medical College & Hospital, Chiplūn, Maharashtra
  - Fortis Hospitals Kalyan, Kalyān, Maharashtra
  - Sir H N Reliance Foundation Hospital, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - S L Raheja Hospital, Mumbai, Maharashtra
  - P.D.Hinduja National Hospital and M.R.C., Mumbai, Maharashtra
  - Bombay Hospital Institute of Medical Sciences, Mumbai, Maharashtra
  - Breach Candy Hospital, Mumbai, Maharashtra
  - Jaslok Hospital, Mumbai, Maharashtra
  - Lilavati Hospital and Research Centre, Mumbai, Maharashtra
  - Nanavati Hospital, Mumbai, Maharashtra
  - Dr. L. H. Hiranandani Hospital, Mumbai, Maharashtra
  - Suretech Hospital, Nagpur, Maharashtra
  - Criticare Hospital & Reaserch Institute, Nagpur, Maharashtra
  - Meditrina Institute of Medical Sciences, Nagpur, Maharashtra
  - Apollo Hospitals, Nashik, Maharashtra
  - Ashoka Medicover hospital, Nashik, Maharashtra
  - Apollo Hospitals, Navi Mumbai, Maharashtra
  - Terna Speciality Hospital and Research Centre, Nerul, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Galaxy care hospital, Pune, Maharashtra
  - Sanjeevan Hospital, Pune, Maharashtra
  - Niramaya Hospital, Pune, Maharashtra
  - Ruby Hall Clinic Wanowrie, Pune, Maharashtra
  - Bharati Vidyapeeth (Deemed to be) University Medical College, Pune, Maharashtra
  - Balwant institute of neurosurgery and intensive trauma care, Solapur, Maharashtra
  - Narayana Super Speciality Hospital, Gurgaon, National Capital Territory of Delhi
  - Nayati Medecity, Mathura, National Capital Territory of Delhi
  - Pushpawati Singhania Research Institute, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - BLK Superspeciality Hospital, New Delhi, National Capital Territory of Delhi
  - Vikash Multispecialty Hospital, Bargarh, Odisha
  - Ims & Sum Hospital, Bhubaneswar, Odisha
  - Apollo Hospitals, Bhubaneswar, Odisha
  - AMRI Hospital, Bhubaneswar, Odisha
  - Ashwini Hospital, Cuttack, Odisha
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - MICU, Deep Hospital, Ludhiana, Punjab
  - Fortis Hospital, Mohali, Punjab
  - Kothari Medical and Research Institute, Bikaner, Rajasthan
  - Santokba Durlabhji Memorial Hospital, Jaipur, Rajasthan
  - Eternal Hospital, Jaipur, Rajasthan
  - JNU Institue of Medical Sciences and Reserach Center, Jaipur, Rajasthan
  - Shubh Hospital, Jaipur, Rajasthan
  - Apollo Hospitals, Chennai, Tamil Nadu
  - Billroth hospital, Chennai, Tamil Nadu
  - Saveetha Medical College and Hospital, Chennai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu
  - vsunshine hospitals, Gachibowli, Hyderabad, Telangana
  - Thumbay Hospital, Hyderabad, Telangana
  - Continental Hospitals, Hyderabad, Telangana
  - Basavatarakam Indo American Cancer Hospital and Research Institute, Hyderabad, Telangana
  - Century Super Specialty Hospital, Hyderabad, Telangana
  - Virinchi Hospital, Hyderabad, Telangana
  - Care Hospital Banjara Hills, Hyderabad, Telangana
  - Pushpanjali Hospital, Agra, Uttar Pradesh
  - Synergy plush hospital, Agra, Uttar Pradesh
  - Medical ICU, Bareilly, Uttar Pradesh
  - Shri Ram Murti Smarak Institute of Medical Sciences, Bareilly, Uttar Pradesh
  - Fortis Hospital, Noida, Uttar Pradesh
  - Jaypee Hospital, Noida, Uttar Pradesh
  - Institute of Medical Sciences, Varanasi, Uttar Pradesh
  - Max Superspeciality Hospital, Dehradun, Uttarakhand
  - Iq City Medical College and Narayana Multi-Specialty Hospital, Durgapur, West Bengal
  - Apollo Gleneagles Hospital, Kolkata, West Bengal
  - Peerless Hospital, Kolkata, West Bengal
  - AMRI Hospitals Salt Lake, Kolkata, West Bengal
  - Amri Hospitals, Kolkata, West Bengal
  - Medica Superspecialty Hospital, Kolkata, West Bengal
  - Fortis, Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Divatia JV, Amin PR, Ramakrishnan N, Kapadia FN, Todi S, Sahu S, Govil D, Chawla R, Kulkarni AP, Samavedam S, Jani CK, Rungta N, Samaddar DP, Mehta S, Venkataraman R, Hegde A, Bande BD, Dhanuka S, Singh V, Tewari R, Zirpe K, Sathe P; INDICAPS Study Investigators. Intensive Care in India: The Indian Intensive Care Case Mix and Practice Patterns Study. Indian J Crit Care Med. 2016 Apr;20(4):216-25. doi: 10.4103/0972-5229.180042. PMID 27186054
- [Derived] Divatia JV, Mehta Y, Govil D, Zirpe K, Amin PR, Ramakrishnan N, Kapadia FN, Sircar M, Sahu S, Bhattacharya PK, Myatra SN, Samavedam S, Dixit S, Pande RK, Mehta SN, Venkataraman R, Bajan K, Kumar V, Harne R, Thakur L, Rathod D, Sathe P, Gurav S, D'Silva C, Pasha SA, Todi SK; the INDICAPS-II investigators. Intensive Care in India in 2018-2019: The Second Indian Intensive Care Case Mix and Practice Patterns Study. Indian J Crit Care Med. 2021 Oct;25(10):1093-1107. doi: 10.5005/jp-journals-10071-23965. PMID 34916740

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients: All patients present in the ICU on the study days were included in the study. Data were recorded for all patients present in the ICU during the 24 hours starting from 08.00 a.m. on the study day to 08.00 a.m. the next day. Neonatal and pediatric ICUs were not included. There were no other exclusion criteria.
Period: Overall Study
Arm/Group | Patients
Started | 5094
Completed | 4669
Not Completed | 425

BASELINE CHARACTERISTICS:
Groups:
- Single Cohort: All patients > 15 years of age present in the intensive care unit on the study days
Arm/Group | Single Cohort
Number analyzed (Participants) | 4669
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1696
  Male | 2973
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Asian (Indian) ethnicity 4669: Hispanic or Latino | 0
  Asian (Indian) ethnicity 4669: Not Hispanic or Latino | 0
  Asian (Indian) ethnicity 4669: Unknown or Not Reported | 4669
Region of Enrollment [Number; unit: participants]
  India | 4669
Age > 15 years [Count of Participants; unit: Participants] | 4669

OUTCOME MEASURES:

1. Primary Outcome: ICU Mortality
Description: Number of patients who died in the ICU, as well as those terminally discharged from the ICU
Time Frame: 30 days from the study day
Measure: Count of Participants; unit: Participants
Arm/Group | Single Cohort
Number analyzed (Participants) | 4669
Participants | 1092

2. Secondary Outcome: Hospital Mortality
Description: all cause hospital mortality, including those terminally discharged from the ICU
Time Frame: 30 days from the study day
Measure: Count of Participants; unit: Participants
Arm/Group | Single Cohort
Number analyzed (Participants) | 4669
Participants | 1164

3. Secondary Outcome: ICU Length of Stay
Description: length of stay in the intensive care unit
Time Frame: upto 30 days from the study day
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Single Cohort
Number analyzed (Participants) | 4669
days | 6 [3 to 13]

4. Secondary Outcome: Hospital Length of Stay
Description: length of stay in the hospital
Time Frame: upto 30 days from the study day
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Single Cohort
Number analyzed (Participants) | 4669
Days | 12 [7 to 20]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Single Cohort
All-Cause Mortality (participants affected / at risk) | 1164/4669
Serious Adverse Events (participants affected / at risk) | 0/4669
Other Adverse Events (participants affected / at risk) | 0/4669

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT03631927/Prot_000.pdf